CLINICAL TRIAL: NCT05921383
Title: Anorectal Manometry of Patients With Constipation Predominant Irritable Bowel Syndrome
Brief Title: Anorectal Manometry of Patients With Constipation Predominant IBS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Sayed Zaki Bebe, resident doctor, Assiut University
Other Study IDs: Anorectal manometery
Record Dates: First submitted 2023-06-18; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Constipation-predominant Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of The study is to compare between the anorectal manometric profile of patients with functional constipation and patients with constipation predominant irritabe bowel syndrome

DETAILED DESCRIPTION:
Chronic constipation (CC) is a common medical problem throughout the world [1-3] The global prevalence of CC in the community varies from 11% to 18% [4].

In patients presenting to tertiary care facilities, specific pathophysiological abnormalities like defecatory disorder and slow colonic transit contribute to CC.

CC has a significant burden on the utilization of healthcare resources, including the cost of inpatient and outpatient care, laboratory tests, and diagnostic procedures [5, 6].

CC is characterized by difficulty in passing stools or a low frequency of bowel movements, often accompanied by straining during defecation or a feeling of incomplete evacuation [7, 8].

For western population, CC is defined by Bristol stool form (BSF) I-II, while in Indian patients, addition of type III Bristol stool form increases diagnostic sensitivity [2]. In the ROME IV criteria, it has been suggested that all patients with CC without evidence of structural or metabolic abnormalities to explain symptoms should be considered under the umbrella of functional constipation (FC) [8].

FC is defined as the presence of two or more of the followings during the previous 3 months:

1. Defecatory straining (> 25% of bowel movements)
2. Hard or lumpy stools (> 25% of bowel movements)
3. Feeling of incomplete evacuation (> 25% of bowel movements)
4. Defecatory obstruction (> 25% of bowel movements)
5. Manual maneuvers to facilitate defecation (> 25% of bowel movements)
6. Fewer than three spontaneous complete bowel movements per week. Symptoms must be present for at least 6 months before the diagnosis, and diarrhea must not be present except after using a laxative [8].

Patients with FC should not meet irritable bowel syndrome (IBS) criteria, although bloating may be present. In contrast, patients with irritable bowel syndrome with constipation (IBS-C) have abdominal pain as the predominant symptom along with Bristol stool form types 1 or 2 more than 25% of the times. [8].

Among patients presenting with CC, Indian studies have reported FC to be commoner than IBS-C [9, 10-12].

High-resolution (HR-) anorectal manometry has significant diagnostic value in the assessment of anorectal disorders [13] This study aimed to compare the clinical and anorectal manometry profile of patients with FC and constipation-predominant irritable bowel syndrome

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18- 60 years old .
2. Patients fulfill ROME IV criteria of chronic constipation.

Exclusion Criteria:

* Patient with secondary causes of constipation :-

  1. Thyroid disease
  2. Acute or chronic kidney disease
  3. Acute or Chronic Liver Disease.
  4. Malignancy 5 -Medication 6 -Uncontrolled diabetes mellitus 7 -Inflammatory bowel diseases

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: both males and females between age 18-60 years
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Value of manometry for diagnosis of functional constipation | 1years
  The aim of The study is to compare between the anorectal manometric profile of patients with functional constipation and patients with constipation predominant irritabe bowel syndrome

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chey WD, Kurlander J, Eswaran S. Irritable bowel syndrome: a clinical review. JAMA. 2015 Mar 3;313(9):949-58. doi: 10.1001/jama.2015.0954. PMID 25734736
- See also: Related Info — http://us.search.yahoo.com/search?fr=yhs-invalid&p=pupmed